CLINICAL TRIAL: NCT04276168
Title: Impact of Iron Stores on Wound Healing in Plastic Surgery
Acronym: IRONPLAST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190575
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-02

CONDITIONS: Healing Wound; Iron-deficiency; Surgical Wound
MeSH Terms: conditions — Anemia, Iron-Deficiency; Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In breast reduction surgery, delayed wound healing may increase surgical site infections, cutaneous necrosis and may be related to psychological harm.Some risk factors have been identified : smoking, diabetes, overweight. A normal healing involve cellular and biochemical reactions in which iron plays an important role such as cellular respiration, redox reactions and regulation of genes involved in the cell cycle. This trial will study the relationship between iron stores and postoperative wound healing after bilateral breast reduction surgery in patients without preoperative anaemia.The primary outcome of this trial is the comparison of wound healing at post operative day 15, between patients with and without iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* female
* scheduled bilateral breast reduction surgery
* biological exams with ferritin and transferrin saturation coefficient taken the day before surgery
* No anemia : haemoglobin >=12g/dL (preoperative biological assessment )
* if genetic disease of haemoglobin, haemoglobin between 10 and 12g/dL and no Anaemia by iron deficiency
* absence of clinical inflammatory syndrome (no clinical signs of infection or no fever)
* non-opposition of the patient to participate

Exclusion Criteria:

* Anaemia by iron deficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort of woman who had a scheduled bilateral breast reduction surgery without anemia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of good breast tissue healing on each breast | 15 days after surgery
  Good healing is defined as a score of 0, 1 or 2 on a 16 points-specifc scale. The scale evaluate proportion of disunity for periareolar vertical and horizontal incisions

SECONDARY OUTCOMES:
Evaluation of healing on the 16 points specific scale | 15 days after surgery
Proportion of early complications | up to 15 days after surgery
Proportion of closed drainage orifices | 15 days after surgery
Correlation between serum ferritin levels before surgery and score on the healing scale | 15 days after surgery
Intra-class correlation coefficient for the healing scale | 15 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided